#### Note to File 1

Official Title: A Phase III, Open label, Randomized, Multi-center Study of the Effects of Leukocyte Interleukin, Injection [Multikine] Plus Standard of Care (Surgery + Radiotherapy or Surgery + Concurrent Chemoradiotherapy) in Subjects with Advanced Primary Squamous Cell Carcinoma of the Oral Cavity / Soft Palate Versus Standard of Care Only

NCT Number: NCT01265849

Date: 28 December 2020

### Note to File Statistical Analysis Plan 28-Dec-2020

### Rationale:

The final SAP signed 27-November-2020 states the following; Note: SAP items 5.2 (2) and (3) and 5.4 (2) and (3) need to be fixed (inadvertent text transposition):

#### To Be Corrected:

# Item 1: Swapped Text (Sections 5.2 and 5.4)

# 5.2 Secondary Hypotheses

The following secondary comparisons are also planned:

(2) LRC for Multikine + CIZ + SOC vs. SOC controlling for pre-planned covariates

Ho: h Multikine + CIZ+ SOC / h SOC = 1 vs.

Ha: h Multikine + soc / h soc < 1,

where h Multikine + CIZ+ SOC is the active (Multikine + CIZ + SOC) hazard rate and h soc is the control (SOC) hazard rate for <u>progression free survival</u> time. TCI E (see Section 4.0) is the main interval of interest.

(3) PFS for Multikine + CIZ + SOC vs. SOC controlling for pre-planned covariates

Ho: h Multikine + CIZ+ soc / h soc = 1 vs.

Ha: h Multikine + soc / h soc < 1,

where h  $_{\text{Multikine}}$  + CIZ+ soc is the active (Multikine + CIZ + SOC) hazard rate and h soc is the control (SOC) hazard rate for  $\underline{\textbf{LRC}}$  (loco-regional control) failure time. TCI E (see Section 4.0) is the main interval of interest.

# **5.4 Other Hypotheses**

(2) <u>LRC</u> for Multikine + CIZ + SOC vs. SOC controlling for pre-planned covariates including histopathology markers

Ho: h Multikine + CIZ+ SOC / h SOC = 1 vs.

Ha: h Multikine + soc / h soc < 1,

where h Multikine + CIZ+ SOC is the active (Multikine + CIZ + SOC) hazard rate and h soc is the control (SOC) hazard rate for <u>PFS</u>.

TCI E (see Section 4.0) is the main interval of interest.

(3) <u>PFS</u> for Multikine + CIZ + SOC vs. SOC controlling for pre-planned covariates including histopathology markers

Ho: h Multikine + CIZ+ soc / h soc = 1 vs.

Ha: h Multikine + soc / h soc < 1,

where h Multikine + CIZ+ SOC is the active (Multikine + CIZ + SOC) hazard rate and h soc is the control (SOC) hazard rate for <u>LRC</u>. TCI E (see Section 4.0) is the main interval of interest.

## Item 1 Solution:

### 5.2 Secondary Hypotheses

The following secondary comparisons are also planned:

(2) LRC for Multikine + CIZ + SOC vs. SOC controlling for pre-planned covariates

Ho: h Multikine + CIZ+ SOC / h SOC = 1 vs.

Ha: h Multikine + soc / h soc < 1,

where h Multikine + CIZ+ SOC is the active (Multikine + CIZ + SOC) hazard rate and h soc is the control (SOC) hazard rate for <u>LRC</u> (loco-regional control) time. TCI E (see Section 4.0) is the main interval of interest.

(3) PFS for Multikine + CIZ + SOC vs. SOC controlling for pre-planned covariates

Ho: h Multikine + CIZ+ soc / h soc = 1 vs.

Ha: h Multikine + soc / h soc < 1,

where h Multikine + CIZ+ SOC is the active (Multikine + CIZ + SOC) hazard rate and h soc is the control (SOC) hazard rate for <u>PFS</u> (progression-free survival) time. TCI E (see Section 4.0) is the main interval of interest.

# 5.4 Other Hypotheses

(2)  $\underline{\textbf{LRC}}$  for Multikine + CIZ + SOC vs. SOC controlling for pre-planned covariates including histopathology markers

Ho: h Multikine + CIZ+ soc / h soc = 1 vs.

Ha: h Multikine + soc / h soc < 1,

where h  $_{\text{Multikine}}$  + CIZ+ SOC is the active (Multikine + CIZ + SOC) hazard rate and h soc is the control (SOC) hazard rate for  $\underline{\textbf{LRC}}$ . TCI E (see Section 4.0) is the main interval of interest.

(3) **PFS** for Multikine + CIZ + SOC vs. SOC controlling for pre-planned covariates including histopathology markers

Ho: h Multikine + CIZ+ SOC / h SOC = 1 vs.

Ha: h Multikine + soc / h soc < 1,

where h Multikine + CIZ+ SOC is the active (Multikine + CIZ + SOC) hazard rate and h soc is the control (SOC) hazard rate for PFS. TCI E (see Section 4.0) is the main interval of interest.

# Item 2: Infeasible DDT Response Analyses (Section 11.1)

In this study, given the disease stage (III and IVa), a blinded review indicated that >90% of study subjects had surgery and that >90% did not have measurable or evaluable disease following surgery. Thus, there will not be sufficient numbers of subjects to be able to be assessed for partial or complete response following subsequent disease-directed treatment (DDT) with which to conduct such analyses, based on the limited capacity of residual disease to be assessed by either measurement or imaging.

#### Item 2 Solution:

Drop the following table and figure series involving DDT response stratification:

- Table Series 14.2.1.1.7
- Table Series 14.2.2.1.5
- Table Series 14.2.3.1.5
- Figure Series 14.2.1.1.8.

# Signatures:

Naping Cai Yaping Cai

29 Dec 2020 13:36:033+0000

REASON: I approve this document 5847fe6f-1cee-4c47-ac55-feff592129f2

> Yaping Cai ICON plc

Phil Lavin

29 Dec 2020 13:55:036+0000

REASON: I approve this document as author.

81797106-ad47-4969-9923-72071d5c68a9

Philip Lavin PhD, FASA, FRAPS Lavin Consulting LLC (CEL-SCI Statistical Consultant)

**Eyal 7alor** Eyal Talor 29 Dec 2020 13:43:027+0000

REASON: I approve this document 5a7c1b19-989b-4b38-8dd9-45225e5fa404

Eyal Talor PhD **CEL-SCI Corp** 

John Cipriano

John Cipriano

29 Dec 2020 15:01:059+0000

REASON: I approve this document 1ab20719-df7a-48a9-9eff-f62f73358e01

John Cipriano CEL-SCI Corp